CLINICAL TRIAL: NCT04945473
Title: Assessment of the Impact of Endoscopic Gastric Revision by Application of Additional Sutures on Weight Loss After Endoscopic Sleeve Gastroplasty in Obese Patients
Brief Title: Gastric Recalibration After Endoscopic Sleeve Gastroplasty
Acronym: ESG-IRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20-006
Record Dates: First submitted 2021-06-08; First posted 2021-06-30 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Morbid Obesity
Keywords: obesity; Endoscopy; ESG; Gastric emptying; Revision procedure
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Revision (Experimental): BMI≥30 or total weight loss (TBWL) < 10% and relaxation of gastric tubulisation at 6 months after ESG.
  Additional stitches will be placed during the follow-up gastroscopy at 6 months.
  Interventions: Procedure: Endoscopic placement of additional sutures
- Without revision (No Intervention): The control gastroscopy will be performed without any additional procedure (no additional stitches).

INTERVENTIONS:
Procedure: Endoscopic placement of additional sutures — A new endoscopic suture will be performed in case of a BMI≥30 or total weight loss (TBWL) less than 10%, and relaxation of gastric tubulization during the regular endoscopic follow-up after 6 months from the ESG. The same endoscopic suture technique of the primary ESG will be applied.
  Arms: Revision

SUMMARY:
Endoscopic sleeve gastroplasty (ESG) is a technique used for bariatric surgery, with results comparable to conventional surgery, in order to treat morbid obesity. It has also less risks of complications, and it is not an irreversible technique. It can be repeated overtime, regarding the evolution of the gastroplasty. There is little data in the literature on the effectiveness of endoscopic "revision". This study will assess the benefits and costs of a revision during the follow-up endoscopy.

DETAILED DESCRIPTION:
Obesity is a health dilemma with an increased risk of premature death. Bariatric surgery is considered to be the most effective and durable treatment for morbid obesity as compared to other available options. However, only the most severe cases, namely class III or class II patients with obesity-related comorbidities fit the criteria for bariatric surgical interventions and are offered these options. Endoscopic sleeve gastroplasty (ESG) is a restrictive procedure based on the tubulization and shortening of the stomach, achieved by means of multiple full-thickness sutures applied endoscopically. ESG offers the possibility to obtain results (weight loss, improvement of comorbidities and quality of life) comparable to conventional surgery while reducing the risk of complications. One of the major advantages of this technique is that it does not make irreversible changes to gastric anatomy and function and can be repeated overtime if needed placing additional sutures. ESG appearance might be subject to changes overtime. In fact, depending on the sutures' integrity, the gastroplasty can be regarded as tight, partially open or completely open. Very little data currently exists in the literature on the effectiveness of endoscopic "revision" with the placement of additional sutures on weight loss and its impact on co-morbidities. In order to objectively assess the benefits and costs of a revision during the follow-up endoscopy patients who present a TWL <10% or a BMI greater than 30 at 6 months from the primary ESG, will be randomized into 2 groups: a "Revision" group in which a revision will be performed systematically in the event of suture disruption at the control EGD, and a "Control" group which will only benefit of a control endoscopy regardless of the state of the gastroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75
* Patients with morbid obesity (BMI≥ 30 with comorbidities or> 40)
* Patients with obesity for more than 2 years
* Failure of medical treatment of obesity
* Patients who may benefit from general anaesthesia
* Patient able to participate in all aspects of the study and that agree to comply with all study requirements, for the duration of the study. This includes the availability of reliable transportation and sufficient time to attend all follow-up visits.
* Patient able to fully understand the study and ready to give consent to participate to the study.
* Patient affiliated to the French social security system

Exclusion Criteria:

* Patient with a contraindication to perform an ESG
* Patient with a history of previous bariatric, gastric or esophageal surgery.
* Patient who initiated medical therapy within the last 3 months, with evidence of weight gain.
* Patient with an uncontrolled, poorly controlled, or suspected history of eating disorders or psychiatric illness.
* Patient with unstable and precarious state of health, as determined and assessed by the investigator.
* Patient who is pregnant, breastfeeding or of childbearing age and without effective contraception.
* Patient in exclusion period (determined by a previous or ongoing study)
* Patient under legal protection
* Patient under guardianship or curatorship
* Patients with a BMI less than 30 at 6 months after ESG. These patients will not be candidate for revision regardless of the randomization group.
* Patients with a contraindication to MRI may be included in the study and will follow the "No Imaging" study design.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Total weight loss (TWL) | 3, 6, 12, 18 and 24 months after the ESG
  The primary endpoint is the assessment of weight evolution in terms of total weight loss (TWL) between the two randomized groups ("Control" vs. "Review"). The evolution of the TWL will be assessed at 3, 6, 12 ,18 and 24 months after the ESG.

SECONDARY OUTCOMES:
Excess weight loss (EWL) | The data will be collected at the follow-up consultation, specifically at 3, 6, 12, 18 and 24 months after the ESG
  Evaluation of weight loss in terms of excess body weight evolution (EWL) between the two randomized groups ("Control" vs. "Review"). The evolution of the EWL will be assessed at 3, 6, 12 ,18 and 24 months after the ESG.
Body mass index (BMI) | The data will be collected at the follow-up consultation, specifically at 3, 6, 12, 18 and 24 months after the ESG
  Evaluation of the weight loss in terms of body mass index (BMI) between the two randomized groups. The evolution of the BMI will be assessed at 3, 6, 12 ,18 and 24 months after the ESG.
Self-esteem and activities evaluation | The data will be collected at the follow-up consultation, specifically at 3, 6, 12, 18 and 24 months after the ESG
  Assessment of the self-esteem and activities before and after the ESG, using the Moorehead-Ardelt quality of life questionnaire II. Score range from -3.0 to 3.0.
  * Score from -3.0 to -2.1: very poor quality of life
  * Score from -2.0 to -1.1: poor quality of life
  * Score from -1.0 to 1.0: fair quality of life
  * Score from 1.1 to 2.0: good quality of life
  * Score from 2.1 to 3.0: very good quality of life. The evolution of will be assessed at 3, 6, 12 ,18 and 24 months after the ESG.
Gastrointestinal quality of life evaluation | The data will be collected at the follow-up consultation, specifically at 3, 6, 12, 18 and 24 months after the ESG
  Assessment of the gastrointestinal quality of life before and after the ESG, using GIQLI (GastroIntestinal Quality of Life Index) questionnaire. There are 36 questions, each ranged from 0 to 4. A global score >125 is considered as normal. The evolution of the gastrointestinal quality of life will be assessed at 3, 6, 12 ,18 and 24 months after the ESG.
Comorbidity evolution | The data will be collected at the follow-up consultation, specifically at 3, 6, 12, 18 and 24 months after the ESG
  Assessment of comorbidities by comparing the evolution of comorbidities (hypertension, diabetes, sleep apnea syndrome, GERD with the questionnaire "GERD-Health Related Quality of Life Questionnaire GERD-HRQL", knee osteoarthritis) before and after the ESG. GERD-HRQL questionnaire contains 16 questions, ranged from 0 to 5. The higher the score is, the more important the gastroesophageal reflux is. The evolution of comorbidities will be assessed at 3, 6, 12 ,18 and 24 months after the ESG.
Gastric Emptying evaluation | The data will be collected before and 7 months after the ESG
  Evaluation of gastric volume and emptying changes before and after ESG. The evaluation will be carried out performing a dynamic MRI before and 7 months after ESG. Dynamic MRI changes will be put in correlation with weight modifications (TWL, EWL and BMI).
Gastric Emptying evaluation | The data will be collected before and 7 months after the ESG
  Evaluation of gastric volume and emptying changes before and after ESG. The evaluation will be carried out performing a dynamic MRI before and 7 months after ESG. Dynamic MRI changes will be put in correlation with changes in secretion of intestinal hormones and glycemic profile (blood sugar, HbA1c, insulin, ghrelin, C-peptide, GLP-1 and Glucagon).
Gastric Emptying evaluation | The data will be collected before and 7 months after the ESG
  Evaluation of changes in gastric volume and gastric emptying comparing the results obtained by dynamic MRI between the two randomized groups ("Control" vs. "Revision"), with an additional correlation study of these results with weight loss: total weight lost (TWL%), excess weight loss (EWL%) and change in BMI. The data will be collected before ESG, and at 3, 6, 12, 18 and 24 months after ESG
Gastric Emptying evaluation | The data will be collected before and 7 months after the ESG
  Evaluation of changes in gastric volume and gastric emptying comparing the results obtained by dynamic MRI between the two randomized groups ("Control" vs. "Revision"), with an additional correlation study of these results with changes in secretion of intestinal hormones and glycemic profile (blood sugar, HbA1c, insulin, ghrelin, C-peptide, GLP-1 and Glucagon). The data will be collected before and 7 months after the ESG.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana PERRETTA, MD, PHD, Principal Investigator — Service de chirurgie digestive et endocrinienne, NHC, Strasbourg
Locations (1):
- Service de chirurgie digestive et endocrinienne, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willett WC, Dietz WH, Colditz GA. Guidelines for healthy weight. N Engl J Med. 1999 Aug 5;341(6):427-34. doi: 10.1056/NEJM199908053410607. No abstract available. PMID 10432328
- [Background] Sharaiha RZ, Kedia P, Kumta N, DeFilippis EM, Gaidhane M, Shukla A, Aronne LJ, Kahaleh M. Initial experience with endoscopic sleeve gastroplasty: technical success and reproducibility in the bariatric population. Endoscopy. 2015 Feb;47(2):164-6. doi: 10.1055/s-0034-1390773. Epub 2014 Nov 7. PMID 25380510
- [Background] Lopez-Nava G, Galvao M, Bautista-Castano I, Fernandez-Corbelle JP, Trell M. Endoscopic sleeve gastroplasty with 1-year follow-up: factors predictive of success. Endosc Int Open. 2016 Feb;4(2):E222-7. doi: 10.1055/s-0041-110771. Epub 2016 Jan 15. PMID 26878054
- [Background] Lopez-Nava G, Galvao MP, Bautista-Castano I, Jimenez-Banos A, Fernandez-Corbelle JP. Endoscopic Sleeve Gastroplasty: How I Do It? Obes Surg. 2015 Aug;25(8):1534-8. doi: 10.1007/s11695-015-1714-7. PMID 26003549
- [Background] Lopez-Nava G, Galvao MP, da Bautista-Castano I, Jimenez A, De Grado T, Fernandez-Corbelle JP. Endoscopic sleeve gastroplasty for the treatment of obesity. Endoscopy. 2015 May;47(5):449-52. doi: 10.1055/s-0034-1390766. Epub 2014 Nov 7. PMID 25380508
- [Background] Abu Dayyeh BK, Rajan E, Gostout CJ. Endoscopic sleeve gastroplasty: a potential endoscopic alternative to surgical sleeve gastrectomy for treatment of obesity. Gastrointest Endosc. 2013 Sep;78(3):530-5. doi: 10.1016/j.gie.2013.04.197. Epub 2013 May 24. PMID 23711556